CLINICAL TRIAL: NCT01580111
Title: Effect of Blood Storage Age on the Resolution of Lactic Acidosis in Children With Severe Malarial Anemia at Mulago Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makerere University (Other)
Responsible Party: Principal Investigator, Faculty of Medicine, Teaching Assistant, Makerere University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AD-001
Record Dates: First submitted 2012-04-17; First posted 2012-04-18 (Estimated); Last update posted 2012-04-18 (Estimated); Status verified 2012-04

CONDITIONS: Compare Blood Age for Transfusion
Keywords: Blood; Storage; Age; Transfusion; Lactic acidosis
MeSH Terms: conditions — Acidosis, Lactic | interventions — Blood Transfusion

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Short storage (Experimental): Short storage arm: Will receive blood (Packed red blood cells) of 1 (one) to 10 (ten) days in storage.
  Interventions: Biological: Blood transfusion
- Long storage arm (Active Comparator): Will be transfused with blood ( packed red cells) of storage age 21- 35 days.
  Interventions: Biological: Blood transfusion

INTERVENTIONS:
Biological: Blood transfusion — The short storage arm; children were transfused with packed red cells of storage age 1-10 days; while for the Long storage arm; were transfused with packed red cells of 21- 35 days in storage.

SUMMARY:
In resolving lactic acidosis among children with severe malarial anemia, there is no difference between those transfused with blood of longer storage compared to shorter storage age

DETAILED DESCRIPTION:
Objective of the study is to evaluate the effect of blood storage age on resolution of lactic acidosis in children with severe malarial anemia.

Methods:

Children aged 6 - 59 months admitted to ACU with Severe Malarial Anemia (Hb <5g/dl) and Lactic Acidosis (blood lactate >5 mmol /l), will be randomly assigned to receive either blood of shorter storage age (<10 days) or longer storage age (21 -35 days) by gravity infusion as is the routine practice. 37 patients will be enrolled in each study arm. Physiological measurements namely blood lactate, oxygen saturation, Hemoglobin, Blood pressure, respiratory rate and pulse rate will be taken at baseline, during and after transfusion. The two groups will be compared. The primary outcome variable will be the proportion of children whose lactic acidosis resolves after 4 hrs of transfusion. 24hr mortality will be our secondary outcome.

ELIGIBILITY:
Inclusion Criteria:Children aged 6 - 59 months admitted at Acute care Unit - Mulago hospital with;

1. A positive B/S for malaria
2. Severe anemia ( Hb ≤ 5 g/dl) and
3. Lactic Acidosis (Blood lactate ≥ 5 mmol/l)
4. Written informed consent from the caretaker.

Exclusion Criteria:

1. Children undergoing transfusion with blood products other than packed cells.
2. Children with known or concurrent cardiac disease.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2010-12; Primary Completion 2011-08 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Effect of blood storage age on the resolution of lactic acidosis in children with severe malarial anemia at Mulago hospital | 4hrs
  The proportion of transfused patients who resolve lactic acidosis within 4 hours of transfusion

SECONDARY OUTCOMES:
Effect of blood storage age on the resolution of lactic acidosis in children with severe malarial anemia at Mulago hospital | 24 HRS
  proportion of children who die within 24 hrs.

CONTACTS AND LOCATIONS:
Overall Officials: AGGREY DHABANGI, MBChB, M.Med, Principal Investigator — Makerere University
Locations (1):
- Mulago Hospital, Kampala, Uganda, Uganda

REFERENCES:
- [Derived] Dhabangi A, Mworozi E, Lubega IR, Cserti-Gazdewich CM, Maganda A, Dzik WH. The effect of blood storage age on treatment of lactic acidosis by transfusion in children with severe malarial anaemia: a pilot, randomized, controlled trial. Malar J. 2013 Feb 6;12:55. doi: 10.1186/1475-2875-12-55. PMID 23388470